CLINICAL TRIAL: NCT01321658
Title: Geriatric Intervention in Elderly Surgical Patients With Colorectal Cancer - a Randomized, Controlled Trial.
Brief Title: Geriatric Intervention in Frail Elderly Patients With Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Cancer Society (Other); University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Torgeir Bruun Wyller, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010/1634
Record Dates: First submitted 2011-03-18; First posted 2011-03-23 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Colorectal Neoplasms
Keywords: Geriatric Assessment; Perioperative Care; Colorectal Neoplasms; Frail Elderly
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Geriatric intervention (Experimental)
  Interventions: Other: Geriatric intervention
- Control (No Intervention)

INTERVENTIONS:
Other: Geriatric intervention — A comprehensive geriatric assessment (CGA), focusing on co-morbidity, medication, cognitive status, depression, nutritional status and physical status is performed. The intervention is individualized according to the results of the CGA.
  Arms: Geriatric intervention

SUMMARY:
This is a randomized, controlled trial on frail elderly patients (aged 65+) with colorectal cancer. The patients will be randomized into two groups. The control group will receive standard surgical treatment. The intervention group will in addition go through a preoperative comprehensive geriatric assessment. The assessment will include evaluation of co-morbidity and medication, social status, nutritional status, cognition, depression and physical performance. This assessment will form basis of an individualized perioperative intervention.

The main aim of the study is to see if the number of postoperative complications in this group can be reduced by a perioperative geriatric intervention. A study of inflammation markers in serum will also be performed, with focus on identifying potential biological frailty markers.

ELIGIBILITY:
Inclusion Criteria:

* Age 65+
* Elective surgery for colorectal cancer
* Frail

Exclusion Criteria:

* Acute surgery
* Not able to consent
* Does not consent with registration

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 122 (Actual)
Dates: Start 2011-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 30 days after surgery

SECONDARY OUTCOMES:
Reoperation | 30 days after surgery
  Number of patients in need of any operation within thirty days after the operation for colorectal cancer.
Readmission | 30 days after surgery
  Number of patients being readmitted to hospital within 30 days after operation for colorectal surgery.
Length of hospital stay | 30 days after surgery
Survival | 3 months after surgery
Quality of life | 3 months after surgery
Living at home or in institution | 3 months after surgery
  Number of patients living at home, with or without formal help, and number of patients living in nursing homes 3 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Torgeir B Wyller, Dr.med, Study Chair — Geriatric dept., Oslo University hospital
Locations (1):
- Dept of gastrointestinal surgery, Oslo University Hospital, Oslo, Norway